CLINICAL TRIAL: NCT01494064
Title: Monitoring of Encephalopathy in Cirrhotic Patients Admitted in Intensive Care Unit : Standardization of Critical Care Nursing
Brief Title: Monitoring of Encephalopathy in Cirrhotic Patients Admitted in Intensive Care
Acronym: STANDAREA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: RCPHRI1018/2
Record Dates: First submitted 2011-12-09; First posted 2011-12-16 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Hepatic Encephalopathy; Liver Cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective: Included patients have been no specific nursing practice.
- Prospective: Standardization of nursing supervision of included patients using a grid of appropriate surveillance for the prevention of complications in the ICU

SUMMARY:
This study seeks to assess the impact of the standardization of nursing supervision of patients with hepatic encephalopathy using a grid of appropriate surveillance for the prevention of complications in the ICU.

DETAILED DESCRIPTION:
As part of improving the quality of care, the paramedic team has developed an evaluation grid quantitative parameters of the early warning score, the Glasgow Coma Score modified and signs suggestive of hepatic encephalopathy.A course of action was later formalized as a function of score when using the grid monitoring.

The aim of the study is to demonstrate that the standardization of monitoring by a quantitative evaluation grid reduces the complications of hepatic encephalopathy. For this, investigator's team will study a before / after standardization by comparing two groups of patients, ICU liver - digestive BEAUJON hospital, and suffering from hepatic encephalopathy associated with liver cirrhosis and therapeutic care project formalized. For the first group have been no specific nursing practice, investigator's team will take a retrospective study. For the second group have been monitoring a standard, investigator's team will take a prospective study.

The total number of patients in each group will be 121 a total of 242. The frequency of pneumonia is the primary outcome. Secondary endpoints were the occurrence of ventilatory disorders, the presence of shock and premature death of the patient during his hospitalization. investigator's team will compare the frequency of occurrence of these complications in both groups.

Data will be collected using a questionnaire based on information from the software and GILDAE DXCARE.

The prospective study will last 26 months. For the retrospective study, the MSI will publish a list of all patients meeting the inclusion criteria and ICU liver - digestive in the 26 months preceding the start of the study.

The interest of this work is to formalize an objective tool for assessing hepatic encephalopathy and improve communication among caregivers.

ELIGIBILITY:
INCLUSION CRITERIA :

* Hepatic encephalopathy
* Liver cirrhosis
* Treatment plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients in Beaujon Hospital as diagnasotic with hepatic encephalopathy and liver cirrhosis and lice which a treatment plan is formalized
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
rate of inhalation pneumonia | 26 months

SECONDARY OUTCOMES:
occurrence of ventilatory disorders | 26 months
presence of shock and premature death of the patient. | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Villard, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Beaujon, Clichy, France